CLINICAL TRIAL: NCT01471496
Title: Prophylactic Injection Therapy Reduces Recurrent Bleeding Rate In Forrest Type IIb Duodenal Ulcer Bleeding
Brief Title: Prophylactic Injection Therapy Reduces Recurrent Bleeding In Forrest Type IIb Duodenal Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: konuk-001
Record Dates: First submitted 2011-11-01; First posted 2011-11-15 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Duodenal Ulcer Bleeding
Keywords: duodenal ulcer; upper gastrointestinal system bleeding; injection therapy
MeSH Terms: conditions — Duodenal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prophylactic injection therapy group (Experimental): In addition to medical therapy which included 2x 30 mg Pantoprazole and intravenous fluids this group of the patients recieved injection therapy.
  Interventions: Procedure: prophylactic injection therapy
- control group (No Intervention): This group of the patients recieved medical therapy only.

INTERVENTIONS:
Procedure: prophylactic injection therapy — Standard application of endoscopic injection therapy as it is used for actively bleeding ulcers, 10 ml of serum saline with 1/10000 epinephrine is submucosally injected to the four quadrants of the ulcer margins.
  Other Names: prophylactic sclerotherapy
  Arms: prophylactic injection therapy group

SUMMARY:
The purpose of this study is to determine whether prophylactic injection therapy reduces recurrent bleeding rate for duodenal ulcers which has the endoscopic stigmata of recent bleeding.

DETAILED DESCRIPTION:
The benefit of endoscopic therapy in ulcers with adherent clots on their surface is still uncertain. A prophylactic injection therapy may reduce the recurrent bleeding rate at this group of patients having this endoscopic stigma of recent bleeding. This type of ulcers are named as type IIb duodenal ulcers according to Forrest's classification, They cary the risk of bleeding recurrence up to 36 percent and as it is reported previously there may be a 12 fold increasement in morbidity and mortality in such cases. A prophylactic endoscopic injection therapy may reduce the risk of recurrent bleeding in this group of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic diagnose of Forrest type 2b duodenal ulcer.

Exclusion Criteria:

* Patients at whom the onset of Upper Gastrointestinal system bleeding symptoms exceeded 24 hours at index endoscopy.
* Patients having hemodynamic instability: systolic blood pressure below 90 mm/hg, heart rate above 110/min
* Demonstration of hemoglobin fall more than 2 g/dl in two hours.
* Patients with coexisting ulcers elsewhere than in duodenum.
* Patients under anticoagulant therapy other than Aspirin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically definitive recurrent bleeding confirmed by upper gastrointestinal system endoscopy or surgery. | within first two days after index endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Osman Z Öner, MD, Principal Investigator — Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Department of General Surgery, Istanbul, Turkey
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Department of General Surgery, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Cheung FK, Lau JY. Management of massive peptic ulcer bleeding. Gastroenterol Clin North Am. 2009 Jun;38(2):231-43. doi: 10.1016/j.gtc.2009.03.003. PMID 19446256
- [Background] Enestvedt BK, Gralnek IM, Mattek N, Lieberman DA, Eisen G. An evaluation of endoscopic indications and findings related to nonvariceal upper-GI hemorrhage in a large multicenter consortium. Gastrointest Endosc. 2008 Mar;67(3):422-9. doi: 10.1016/j.gie.2007.09.024. Epub 2008 Jan 18. PMID 18206878
- [Background] Yavorski RT, Wong RK, Maydonovitch C, Battin LS, Furnia A, Amundson DE. Analysis of 3,294 cases of upper gastrointestinal bleeding in military medical facilities. Am J Gastroenterol. 1995 Apr;90(4):568-73. PMID 7717312
- [Background] Pilotto A, Maggi S, Noale M, Franceschi M, Parisi G, Crepaldi G; IPOD Investigators. Development and validation of a new questionnaire for the evaluation of upper gastrointestinal symptoms in the elderly population: a multicenter study. J Gerontol A Biol Sci Med Sci. 2010 Feb;65(2):174-8. doi: 10.1093/gerona/glp073. Epub 2009 Jun 15. PMID 19528359
- [Background] Cappell MS, Friedel D. Initial management of acute upper gastrointestinal bleeding: from initial evaluation up to gastrointestinal endoscopy. Med Clin North Am. 2008 May;92(3):491-509, xi. doi: 10.1016/j.mcna.2008.01.005. PMID 18387374
- [Background] Kovacs TO. Management of upper gastrointestinal bleeding. Curr Gastroenterol Rep. 2008 Dec;10(6):535-42. doi: 10.1007/s11894-008-0099-3. PMID 19006607
- [Background] Kubba AK, Palmer KR. Role of endoscopic injection therapy in the treatment of bleeding peptic ulcer. Br J Surg. 1996 Apr;83(4):461-8. doi: 10.1002/bjs.1800830408. PMID 8665233
- [Background] Chung SC, Leung JW, Leung FW. Effect of submucosal epinephrine injection on local gastric blood flow. A study using laser Doppler flowmetry and reflectance spectrophotometry. Dig Dis Sci. 1990 Aug;35(8):1008-11. doi: 10.1007/BF01537250. PMID 2384031
- [Background] Calvet X, Vergara M, Brullet E, Gisbert JP, Campo R. Addition of a second endoscopic treatment following epinephrine injection improves outcome in high-risk bleeding ulcers. Gastroenterology. 2004 Feb;126(2):441-50. doi: 10.1053/j.gastro.2003.11.006. PMID 14762781
- [Background] Green FW Jr, Kaplan MM, Curtis LE, Levine PH. Effect of acid and pepsin on blood coagulation and platelet aggregation. A possible contributor prolonged gastroduodenal mucosal hemorrhage. Gastroenterology. 1978 Jan;74(1):38-43. PMID 21830
- [Background] Heldwein W, Schreiner J, Pedrazzoli J, Lehnert P. Is the Forrest classification a useful tool for planning endoscopic therapy of bleeding peptic ulcers? Endoscopy. 1989 Nov;21(6):258-62. doi: 10.1055/s-2007-1010729. PMID 2693077
- [Background] Ferguson CB, Mitchell RM. Non-variceal upper gastrointestinal bleeding. Ulster Med J. 2006 Jan;75(1):32-9. No abstract available. PMID 16457402
- [Background] Forrest JA, Finlayson ND, Shearman DJ. Endoscopy in gastrointestinal bleeding. Lancet. 1974 Aug 17;2(7877):394-7. doi: 10.1016/s0140-6736(74)91770-x. No abstract available. PMID 4136718
- [Background] Peter S, Wilcox CM. Modern endoscopic therapy of peptic ulcer bleeding. Dig Dis. 2008;26(4):291-9. doi: 10.1159/000177011. Epub 2009 Jan 30. PMID 19188717
- [Background] Armstrong CP, Blower AL. Non-steroidal anti-inflammatory drugs and life threatening complications of peptic ulceration. Gut. 1987 May;28(5):527-32. doi: 10.1136/gut.28.5.527. PMID 3596334
- [Background] Balanzo J, Sainz S, Such J, Espinos JC, Guarner C, Cusso X, Mones J, Vilardell F. Endoscopic hemostasis by local injection of epinephrine and polidocanol in bleeding ulcer. A prospective randomized trial. Endoscopy. 1988 Nov;20(6):289-91. doi: 10.1055/s-2007-1013023. PMID 3068050
- [Background] Buffoli F, Graffeo M, Nicosia F, Gentile C, Cesari P, Rolfi F, Paterlini A. Peptic ulcer bleeding: comparison of two hemostatic procedures. Am J Gastroenterol. 2001 Jan;96(1):89-94. doi: 10.1111/j.1572-0241.2001.03456.x. PMID 11197294
- [Background] Hui WM, Ng MM, Lok AS, Lai CL, Lau YN, Lam SK. A randomized comparative study of laser photocoagulation, heater probe, and bipolar electrocoagulation in the treatment of actively bleeding ulcers. Gastrointest Endosc. 1991 May-Jun;37(3):299-304. doi: 10.1016/s0016-5107(91)70719-0. PMID 2070978
- [Background] Cook DJ, Guyatt GH, Salena BJ, Laine LA. Endoscopic therapy for acute nonvariceal upper gastrointestinal hemorrhage: a meta-analysis. Gastroenterology. 1992 Jan;102(1):139-48. doi: 10.1016/0016-5085(92)91793-4. PMID 1530782
- [Background] Branicki FJ, Coleman SY, Fok PJ, Pritchett CJ, Fan ST, Lai EC, Mok FP, Cheung WL, Lau PW, Tuen HH, et al. Bleeding peptic ulcer: a prospective evaluation of risk factors for rebleeding and mortality. World J Surg. 1990 Mar-Apr;14(2):262-9; discussion 269-70. doi: 10.1007/BF01664889. PMID 2327100
- [Background] Cooper GS, Chak A, Way LE, Hammar PJ, Harper DL, Rosenthal GE. Early endoscopy in upper gastrointestinal hemorrhage: associations with recurrent bleeding, surgery, and length of hospital stay. Gastrointest Endosc. 1999 Feb;49(2):145-52. doi: 10.1016/s0016-5107(99)70478-5. PMID 9925690
- [Background] Laine L, McQuaid KR. Endoscopic therapy for bleeding ulcers: an evidence-based approach based on meta-analyses of randomized controlled trials. Clin Gastroenterol Hepatol. 2009 Jan;7(1):33-47; quiz 1-2. doi: 10.1016/j.cgh.2008.08.016. Epub 2008 Aug 16. PMID 18986845
- [Background] Kahi CJ, Jensen DM, Sung JJ, Bleau BL, Jung HK, Eckert G, Imperiale TF. Endoscopic therapy versus medical therapy for bleeding peptic ulcer with adherent clot: a meta-analysis. Gastroenterology. 2005 Sep;129(3):855-62. doi: 10.1053/j.gastro.2005.06.070. PMID 16143125
- [Background] Marmo R, Rotondano G, Bianco MA, Piscopo R, Prisco A, Cipolletta L. Outcome of endoscopic treatment for peptic ulcer bleeding: Is a second look necessary? A meta-analysis. Gastrointest Endosc. 2003 Jan;57(1):62-7. doi: 10.1067/mge.2003.48. PMID 12518133
- [Background] Laine L, Stein C, Sharma V. A prospective outcome study of patients with clot in an ulcer and the effect of irrigation. Gastrointest Endosc. 1996 Feb;43(2 Pt 1):107-10. doi: 10.1016/s0016-5107(06)80109-4. PMID 8635701